CLINICAL TRIAL: NCT01530724
Title: Effect of Weight-loss Diet Strategies and Exercise on Dynamics of Body Fat Depots and Metabolic Rate
Brief Title: Diet and Body Composition
Acronym: CENTRAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Iris Shai, Iris Shai, RD PhD, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ISF256/09; 256/09 (Other Grant/Funding Number: ISF256/09)
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: abdominal obesity
MeSH Terms: conditions — Obesity; Obesity, Abdominal | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low fat diet (Experimental): Weight-loss diet strategy
  Interventions: Other: Weight-loss diet strategy (+) exercise (PA); Other: weight loss (-) exercise (PA)
- low carb diet (Experimental): Weight-loss diet strategy
  Interventions: Other: Weight-loss diet strategy (+) exercise (PA); Other: weight loss (-) exercise (PA)

INTERVENTIONS:
Other: Weight-loss diet strategy (+) exercise (PA) — Weight-loss diet strategy with a free gym membership; monthly 60-minute educational workshops; 3 sessions of workout per week of mostly aerobic training
Other: weight loss (-) exercise (PA) — Weight-loss diet strategy without exercise

SUMMARY:
The investigators hypothesize that differential dynamics in fat depots in response to two opposing dietary strategies mediate the beneficial metabolic effects during weight loss and regain phases.

ELIGIBILITY:
Inclusion Criteria:

* Elevated waist circumference:

  * Men: > 40 inches (102 cm)
  * Women> 35 inches (88 cm)
* Poor dieters with TG>150mg/dL and high-density-lipoprotein cholesterol [HDL-c] <40 mg/dL for men and <50 mg/dL for women

Exclusion Criteria:

* Pregnant or lactating women
* Serum creatinine LT 2 mg/dl
* Disturbed liver function (LT 3 fold level of ALT and AST enzymes)
* Active cancer
* Individuals who cannot start physical activity in the gym
* Individuals that are highly physically active (more than 4 hours/week)
* Active in other nutritional trial

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
body fat composition | 0, 6,18 months
  changes in body fat (MRI)
obesity | 0, 6, 18 months
  changes in weight
abdominal obesity | 0, 6, 18 months
  changes in waist circumference

SECONDARY OUTCOMES:
Lipid profile | 0, 6, 18 months
  Changes in lipid biomarkers: total cholesterol (mg/dL), triglycerides (mg/dL), HDLc (mg/dL), LDLc (mg/dL) (blood draw)
Glycemic control | 0, 6, 18 months
  Changes in fasting glucose (mg/dL) (blood draw)
Glycemic control | 0, 6, 18 months
  Changes in insulin (μIU/mL) (blood draw)
Inflammatory state | 0, 6, 18 months
  Changes hsCRP (mg/L) (blood draw)
Metabolomic | 0, 6, 18 months
  Changes in sub-lipids (blood draw)
Metabolomic | 0, 6, 18 months
  Changes in sub-proteins ( blood draw)
Liver function (blood biomarkers) | 0, 6, 18 months
  Changes in ALT (U/l), AST (U/l), ALKP (U/I), GGT (U/l) (blood draw)
Genetic signature | baseline
  SNPs (variants) associated with fat distribution and visceral fat (blood draw)
Epigenetics | 0, 6, 18 months
  changes in genes' methylation (blood draw)
Epigenetics | 0, 6, 18 months
  changes in mRNAs (blood draw)

CONTACTS AND LOCATIONS:
Locations (1):
- nuclear research center Negev, Dimona, Israel

REFERENCES:
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Derived] Klein H, Pachter D, Goldberg Toren DT, Kamer O, Alufer L, Ebstein Karamani N, Chassidim Y, Shelef I, Rudich A, Yoel U, Ben-Arie G, Zelicha H, Yaskolka Meir A, Tsaban G, Bartal C, Bluher M, Stumvoll M, Ceglarek U, Isermann B, Qi L, Stampfer MJ, Hu FB, Shai I. How effective is rejoining a long-term weight loss program? The 5- and 10-year MRI-assessed Follow Interventions Trial (FIT) project. BMC Med. 2026 Jan 30. doi: 10.1186/s12916-026-04663-9. Online ahead of print. PMID 41612310
- [Derived] Yaskolka Meir A, Tsaban G, Rinott E, Zelicha H, Schwarzfuchs D, Gepner Y, Rudich A, Shelef I, Bluher M, Stumvoll M, Ceglarek U, Isermann B, Kloting N, Keller M, Kovacs P, Qi L, Wang DD, Liang L, Hu FB, Stampfer MJ, Shai I. Individual response to lifestyle interventions: a pooled analysis of three long-term weight loss trials. Eur J Prev Cardiol. 2025 Nov 11;32(16):1660-1670. doi: 10.1093/eurjpc/zwaf308. PMID 40472282
- [Derived] Klein H, Zelicha H, Yaskolka Meir A, Rinott E, Tsaban G, Kaplan A, Chassidim Y, Gepner Y, Bluher M, Ceglarek U, Isermann B, Stumvoll M, Shelef I, Qi L, Li J, Hu FB, Stampfer MJ, Shai I. Visceral adipose tissue area and proportion provide distinct reflections of cardiometabolic outcomes in weight loss; pooled analysis of MRI-assessed CENTRAL and DIRECT PLUS dietary randomized controlled trials. BMC Med. 2025 Feb 4;23(1):57. doi: 10.1186/s12916-025-03891-9. PMID 39901232
- [Derived] Heianza Y, Krohn K, Yaskolka Meir A, Wang X, Ziesche S, Ceglarek U, Bluher M, Keller M, Kovacs P, Shai I, Qi L. Changes in Circulating miR-375-3p and Improvements in Visceral and Hepatic Fat Contents in Response to Lifestyle Interventions: The CENTRAL Trial. Diabetes Care. 2022 Aug 1;45(8):1911-1913. doi: 10.2337/dc21-2517. PMID 35657082
- [Derived] Heianza Y, Krohn K, Xue Q, Yaskolka Meir A, Ziesche S, Ceglarek U, Bluher M, Keller M, Kovacs P, Shai I, Qi L. Changes in circulating microRNAs-99/100 and reductions of visceral and ectopic fat depots in response to lifestyle interventions: the CENTRAL trial. Am J Clin Nutr. 2022 Jul 6;116(1):165-172. doi: 10.1093/ajcn/nqac070. PMID 35348584
- [Derived] Tsaban G, Bilitzky-Kopit A, Yaskolka Meir A, Zelicha H, Gepner Y, Shelef I, Orr O, Chassidim Y, Sarusi B, Ceglarek U, Stumvoll M, Bluher M, Stampfer MJ, Shai I, Schwarzfuchs D. The Effect of Weight-Loss Interventions on Cervical and Chin Subcutaneous Fat Depots; the CENTRAL Randomized Controlled Trial. Nutrients. 2021 Oct 27;13(11):3827. doi: 10.3390/nu13113827. PMID 34836081
- [Derived] Yaskolka Meir A, Keller M, Muller L, Bernhart SH, Tsaban G, Zelicha H, Rinott E, Kaplan A, Gepner Y, Shelef I, Schwarzfuchs D, Ceglarek U, Stadler P, Bluher M, Stumvoll M, Kovacs P, Shai I. Effects of lifestyle interventions on epigenetic signatures of liver fat: Central randomized controlled trial. Liver Int. 2021 Sep;41(9):2101-2111. doi: 10.1111/liv.14916. Epub 2021 May 28. PMID 33938135
- [Derived] Yaskolka Meir A, Keller M, Bernhart SH, Rinott E, Tsaban G, Zelicha H, Kaplan A, Schwarzfuchs D, Shelef I, Gepner Y, Li J, Lin Y, Bluher M, Ceglarek U, Stumvoll M, Stadler PF, Stampfer MJ, Kovacs P, Liang L, Shai I. Lifestyle weight-loss intervention may attenuate methylation aging: the CENTRAL MRI randomized controlled trial. Clin Epigenetics. 2021 Mar 4;13(1):48. doi: 10.1186/s13148-021-01038-0. PMID 33663610
- [Derived] Gepner Y, Goldstein N, Shelef I, Schwarzfuchs D, Zelicha H, Meir AY, Tsaban G, Grossman E. Dissociation Between Long-term Weight Loss Intervention and Blood Pressure: an 18-month Randomized Controlled Trial. J Gen Intern Med. 2021 Aug;36(8):2300-2306. doi: 10.1007/s11606-021-06655-2. Epub 2021 Feb 25. PMID 33634382
- [Derived] Gepner Y, Shelef I, Komy O, Cohen N, Schwarzfuchs D, Bril N, Rein M, Serfaty D, Kenigsbuch S, Zelicha H, Yaskolka Meir A, Tene L, Bilitzky A, Tsaban G, Chassidim Y, Sarusy B, Ceglarek U, Thiery J, Stumvoll M, Bluher M, Stampfer MJ, Rudich A, Shai I. The beneficial effects of Mediterranean diet over low-fat diet may be mediated by decreasing hepatic fat content. J Hepatol. 2019 Aug;71(2):379-388. doi: 10.1016/j.jhep.2019.04.013. Epub 2019 May 8. PMID 31075323
- [Derived] Tene L, Shelef I, Schwarzfuchs D, Gepner Y, Yaskolka Meir A, Tsaban G, Zelicha H, Bilitzky A, Komy O, Cohen N, Bril N, Rein M, Serfaty D, Kenigsbuch S, Chassidim Y, Sarusy B, Ceglarek U, Stumvoll M, Bluher M, Thiery J, Stampfer MJ, Rudich A, Shai I. The effect of long-term weight-loss intervention strategies on the dynamics of pancreatic-fat and morphology: An MRI RCT study. Clin Nutr ESPEN. 2018 Apr;24:82-89. doi: 10.1016/j.clnesp.2018.01.008. Epub 2018 Feb 6. PMID 29576369
- [Derived] Gepner Y, Shelef I, Schwarzfuchs D, Cohen N, Bril N, Rein M, Tsaban G, Zelicha H, Yaskolka Meir A, Tene L, Sarusy B, Rosen P, Hoffman JR, Stout JR, Thiery J, Ceglarek U, Stumvoll M, Bluher M, Stampfer MJ, Shai I. Intramyocellular triacylglycerol accumulation across weight loss strategies; Sub-study of the CENTRAL trial. PLoS One. 2017 Nov 30;12(11):e0188431. doi: 10.1371/journal.pone.0188431. eCollection 2017. PMID 29190720
- [Derived] Gepner Y, Shelef I, Schwarzfuchs D, Zelicha H, Tene L, Yaskolka Meir A, Tsaban G, Cohen N, Bril N, Rein M, Serfaty D, Kenigsbuch S, Komy O, Wolak A, Chassidim Y, Golan R, Avni-Hassid H, Bilitzky A, Sarusi B, Goshen E, Shemesh E, Henkin Y, Stumvoll M, Bluher M, Thiery J, Ceglarek U, Rudich A, Stampfer MJ, Shai I. Effect of Distinct Lifestyle Interventions on Mobilization of Fat Storage Pools: CENTRAL Magnetic Resonance Imaging Randomized Controlled Trial. Circulation. 2018 Mar 13;137(11):1143-1157. doi: 10.1161/CIRCULATIONAHA.117.030501. Epub 2017 Nov 15. PMID 29142011
- [Derived] Tsaban G, Wolak A, Avni-Hassid H, Gepner Y, Shelef I, Henkin Y, Schwarzfuchs D, Cohen N, Bril N, Rein M, Serfaty D, Kenigsbuch S, Tene L, Zelicha H, Yaskolka-Meir A, Komy O, Bilitzky A, Chassidim Y, Ceglarek U, Stumvoll M, Bluher M, Thiery J, Dicker D, Rudich A, Stampfer MJ, Shai I. Dynamics of intrapericardial and extrapericardial fat tissues during long-term, dietary-induced, moderate weight loss. Am J Clin Nutr. 2017 Oct;106(4):984-995. doi: 10.3945/ajcn.117.157115. Epub 2017 Aug 16. PMID 28814394
- [Derived] Zelicha H, Schwarzfuchs D, Shelef I, Gepner Y, Tsaban G, Tene L, Yaskolka Meir A, Bilitzky A, Komy O, Cohen N, Bril N, Rein M, Serfaty D, Kenigsbuch S, Chassidim Y, Sarusi B, Thiery J, Ceglarek U, Stumvoll M, Bluher M, Haviv YS, Stampfer MJ, Rudich A, Shai I. Changes of renal sinus fat and renal parenchymal fat during an 18-month randomized weight loss trial. Clin Nutr. 2018 Aug;37(4):1145-1153. doi: 10.1016/j.clnu.2017.04.007. Epub 2017 May 2. PMID 28501343